CLINICAL TRIAL: NCT07273487
Title: Nurse Education on Ventilator Waveform and Alarm Management and Its Impact on Patient-Ventilator Asynchrony and Clinical Outcomes in the Pediatric Intensive Care Unit: A Prospective Cluster-Randomized Controlled Quality Improvement Study
Brief Title: Nurse Education to Reduce Patient-Ventilator Asynchrony in the PICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Hasan ağın, Prof.Dr, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025/977
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Patient-Ventilator Asynchrony; Mechanical Ventilation Complication; Nurse Education
MeSH Terms: conditions — Patient-Ventilator Asynchrony

STUDY DESIGN:
Intervention Model Description: Two pediatric intensive care units were randomized as clusters to Education vs Control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): Bedside nurses received a structured multimodal education program on ventilator waveform interpretation, recognition of patient-ventilator asynchrony, and ventilator alarm management. The training included face-to-face sessions, case-based waveform discussions, reference pocket cards, and real-time waveform sharing with an asynchrony review team. Nurses conducted routine waveform checks and communicated suspected asynchrony to physicians; ventilator adjustments were performed only by physicians.
  Interventions: Behavioral: Nurse Education on Ventilator Waveform and Alarm Management
- Control Group (No Intervention): Patients received standard care in accordance with existing mechanical ventilation and alarm management protocols. No nurse-specific training on ventilator waveforms or patient-ventilator asynchrony was provided. Asynchrony was assessed using 24-hour ventilator waveform recordings exported for analysis.

INTERVENTIONS:
Behavioral: Nurse Education on Ventilator Waveform and Alarm Management — A structured multimodal education program delivered to bedside nurses, including face-to-face teaching, case-based ventilator waveform interpretation, recognition of common patient-ventilator asynchrony patterns, ventilator alarm management principles, reference pocket cards, and real-time waveform sharing with an asynchrony review team. Nurses performed routine waveform checks and reported suspected asynchrony to physicians; ventilator adjustments were performed only by physicians.
  Other Names: Ventilator Waveform Training
  Arms: Education Group

SUMMARY:
A prospective cluster-randomized quality improvement trial was conducted to evaluate whether a structured nurse education program on ventilator waveform interpretation and alarm management reduces patient-ventilator asynchrony in the pediatric intensive care unit. Two PICU units within the same hospital were randomized to either an Education group or a Control group. Nurses in the Education group received multimodal training, reference cards, and support for real-time waveform review. The primary outcomes were asynchrony index (%) and ventilator alarm frequency (alarms/day). Secondary outcomes included ventilator days, cumulative sedation dose, withdrawal symptoms, nurse accuracy in identifying asynchrony, and nurse workload.

DETAILED DESCRIPTION:
Patient-ventilator asynchrony (PVA) is common in mechanically ventilated children and is associated with impaired gas exchange, increased sedation exposure, prolonged mechanical ventilation, and higher morbidity. Recognition and management of asynchrony require real-time waveform interpretation, yet bedside nurses' ability to identify it varies widely.

This prospective cluster-randomized quality improvement study was conducted in two pediatric intensive care units within the same tertiary children's hospital. The two PICUs were randomized 1:1 to either the Education group or the Control group. Children aged 1 month to 18 years who required at least 48 hours of invasive mechanical ventilation were eligible.

In the Education group, bedside nurses participated in a structured, multimodal training program including face-to-face teaching, case-based waveform analysis, alarm management principles, and a mobile platform for sharing ventilator screenshots with an asynchrony review team. Reference pocket cards summarizing common asynchrony patterns and recommended responses were provided. Nurses performed routine waveform checks and communicated suspected asynchrony to the clinical team; ventilator settings were changed only by physicians.

The Control group followed the existing standard of care without nurse-specific training. Asynchrony was quantified using 24-hour waveform recordings exported from the ventilator.

Primary outcomes were asynchrony index (%) and total ventilator alarm frequency (alarms per ventilator day). Secondary outcomes included mechanical ventilation duration, cumulative sedation dose (mg/kg), withdrawal symptoms measured using the WAT-1 score, nurse accuracy before and after training, and nurse workload assessed using the NASA-TLX tool.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 18 years
* Admission to the pediatric intensive care unit (PICU)
* Receiving invasive mechanical ventilation for at least 48 hours (expected or actual)
* Managed with ventilators capable of waveform monitoring and data export

Exclusion Criteria:

* Use of continuous neuromuscular blocking agents
* Hemodynamic instability preventing study procedures
* Expected duration of invasive mechanical ventilation < 48 hours
* Lack of informed consent (if applicable per ethics approval)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Asynchrony Index (%) | Within the first 24 hours of invasive mechanical ventilation
  The proportion of asynchronous breaths divided by total breaths, expressed as a percentage. Asynchrony is quantified using 24-hour ventilator waveform recordings.
Ventilator Alarm Frequency (alarms/day) | Within the first 24 hours of invasive mechanical ventilation
  The total number of ventilator alarms per ventilator day, including pressure, volume, and flow-related alarms.

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation (days) | Up to 28 days or until discontinuation of invasive mechanical ventilation, whichever comes first.
  Number of days from initiation of invasive mechanical ventilation to successful extubation or transition to noninvasive ventilation.
Cumulative Sedation Dose (mg/kg) | Up to 28 days or until discontinuation of invasive mechanical ventilation, whichever comes first.
  Total cumulative dose of sedative medications administered during mechanical ventilation, normalized to patient weight.
Nurse Accuracy in Identifying Asynchrony (%) | Within the first 24 hours of invasive mechanical ventilation
  Proportion of correctly identified asynchrony patterns on pre-training and post-training waveform tests.
Withdrawal Severity (WAT-1 Score) | Up to 48 hours after extubation following a period of mechanical ventilation.
  Maximum Withdrawal Assessment Tool-1 (WAT-1) score recorded during mechanical ventilation and weaning.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Prof.Dr., Principal Investigator — Dr. Behcet Uz Children's Hospital
Locations (1):
- Behcet Uz Children's Hospital - Pediatric Intensive Care Unit, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data.